CLINICAL TRIAL: NCT06191419
Title: Human Perception of Odors and Odor Blockers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tim McClintock (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Tim McClintock, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 43123; 1K18DC020155 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Smoking; Smoking Behaviors
Keywords: Odors; Sensory perception; Nicotine addiction; Motivation
MeSH Terms: conditions — Tobacco Smoking; Smoking; Tobacco Use Disorder | interventions — Odorants

STUDY DESIGN:
Intervention Model Description: Each subject experiences and reports on all of the odor blocker and control treatments.
Masking Description: Odor bags are prepared by one staff member and labeled with a code so that other investigators administering tests cannot identify which treatment is being given and inadvertently influence outcomes. The code is not visible to participants. This prevents participants from anticipating the effect of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants that Smoke (Experimental): Each smoker is asked to smell up to 20 samples per session. Samples include controls (clean air, irrelevant odor), blocking odors, cigarette smoke, and cigarette smoke mixed with blocking odors or irrelevant odors.
  Interventions: Other: Odorants

INTERVENTIONS:
Other: Odorants — Each smoker is assigned a CPAP nose mask. Odor sample bags are attached to the mask. Smokers open the valve, inhale once through the nose, close the valve, remove the bag from the mask and report on the odor.

SUMMARY:
The goal of this clinical trial is to determine whether blockers of perception of key odorants in cigarette smoke have any utility in smoking cessation. The main question it aims to answer is:

• Can odor blockers be used to suppress perception of the intensity of cigarette smoke in ways that reduce the ability of the odor of cigarette smoke to increase the urge to smoke.

Participants will be asked to smell up to 20 odor samples per session and report on odor pleasantness and desire to smoke.

DETAILED DESCRIPTION:
The experimental treatments include controls (clean air, irrelevant odor), blocking odors, cigarette smoke odor, and cigarette smoke odor mixed with blocking odors or irrelevant odor. To obtain cigarette smoke odor a 1 inch length of a 1R6F research cigarette is burned to completion in a sealed 5 gallon chamber fitted with septa. Using a syringe fit with a needle and filter, 60 mL aliquots of smoke odor are obtained. These smoke odor aliquots, along with blocking odors, are injected into odor sample bags fit with a septum and a valve that can be attached to the CPAP nose mask worn by each participating smoker. Participants open the valve, inhale once through the nose, close the valve, and then remove the bag from the mask before reporting odor pleasantness and the desire to smoke. A 2 - 3 min wait period is enforced between each odor presentation to prevent odor adaptation and to allow acute motivational effects to subside.

In a testing session a participant sniffs 4 concentrations of a mixture of 2 blocking odors, along with control odor samples. Presentation order is randomized. Each participant is assigned their own CPAP nose mask, and masks are disinfected after use. Participants also provide demographic (age, sex, ethnic and racial background) and smoking history information (cigarettes per day, preferred brand, age at onset, and time since last cigarette).

ELIGIBILITY:
Inclusion Criteria:

* Smoker

Exclusion Criteria:

* Non Smoker
* Self reported inability to smell or taste

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Cigarette Purchase Task | 3 hours (total for all outcome measures)
  The Cigarette Purchase Task (Strickland et al., 2016) requires selecting how much the smoker is willing to spend for a single cigarette (their preferred brand) from a list of 19 amounts ranging from $0.00 (free) to $1,120.
Desire to Smoke | 3 hours (total for all outcome measures)
  A rating of participant's desire to smoke on a scale of 0 - 100, where a higher score indicates increased desire.

SECONDARY OUTCOMES:
Odor pleasantness score | 3 hours (total for all outcome measures)
  Participants complete a forced choice test by scoring whether the odor is pleasant or unpleasant

CONTACTS AND LOCATIONS:
Overall Officials: Timothy McClintock, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06191419/ICF_000.pdf